CLINICAL TRIAL: NCT01825850
Title: A Randomized, Open Label Crossover Study to Investigate the Pharmacokinetic Drug Interactions Between Gemigliptin and Irbesartan in Healthy Male Subjects
Brief Title: Pharmacokinetic Drug Interaction Study Between Gemigliptin and Irbesartan After Oral Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: LG-GBCL001
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — LC15-0444; Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gemigliptin (Experimental): Gemigliptin 50mg q.d. during 7 days
  Interventions: Drug: Gemigliptin
- Irbesartan (Experimental): Irbesartan 300mg q.d. during 7 days
  Interventions: Drug: Irbesartan
- Gemiglitin + Irbesartan (Experimental): Gemigliptin 50mg + Irbesartan 300mg q.d. during 7 days
  Interventions: Drug: Gemigliptin; Drug: Irbesartan

INTERVENTIONS:
Drug: Gemigliptin
  Arms: Gemigliptin; Gemiglitin + Irbesartan
Drug: Irbesartan
  Arms: Gemiglitin + Irbesartan; Irbesartan

SUMMARY:
The objective of the study is to investigate the drug interaction between Gemigliptin and Irbesartan by comparing pharmacokinetics of Gemigliptin and Irbesartan administered concomitantly and each alone in healthy male subjects.

ELIGIBILITY:
* Inclusion Criteria

  * Age between 20 to 45, healthy male subjects (at screening)
  * BMI between 18 - 27 kg/m2 (at screening)
  * Blood pressure SBP 90-140 mmHg, DBP 60-95 mmHg
  * FPG 70-125mg/dL glucose level (at screening)
  * Subject who totally understand the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the
* Exclusion Criteria

  * Subject who has past or present history of any diseases following below.(liver including hepatitis virus carrier, kidney, Neurology,immunology,pulmonary,endocrine,hematooncology,cardiology,mental disorder.)
  * Subject who had GI tract disease that influencable to drug absorption or(ulcer, acute or chronic pancreatitis) surgery.(appendectomy, hernioplasty are not included)
  * Subject who had drug hypersensitivity reaction.(gemigliptin, irbesartan, aspirin, antibiotics)
  * Subject who already admitted in other investigator product in 80 days
  * Subject who had whole blood donation in 60 days, or component blood donation in 30 days or transfusion in 30 days currently

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Cmax,ss | up to 72h post-dose
  To evaluate Cmax,ss of Gemigliptin and Irbesartan
AUCτ,ss | up to 72h post-dose
  To evaluate AUCτ,ss of Gemigliptin and Irbesartan

SECONDARY OUTCOMES:
Cmin,ss | up to 72h post-dose
  To evaluate Cmin,ss of Gemigliptin and Irbesartan
Tmax,ss | up to 72h post-dose
  To evaluate Tmax,ss of Gemigliptin, Irbesartan and LC15-0636 (active metaboilite of Gemigliptin)
Cmax,ss | up to 72h post-dose
  To evaluate Cmax,ss of LC15-0636 (active metaboilite of Gemigliptin)
AUCτ,ss | up to 72h post-dose
  To evaluate AUCτ,ss of LC15-0636(active metabolite of Gemigliptin)
metabolic ratio | up to 72h post-dose
  To evaluate metabolic ratio of LC15-0636(active metabolite of Gemigliptin)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Choi HY, Lim HS, Kim YH, Jeon HS, Kim MJ, Lee SH, Jung JH, Lee YK, Kim HJ, Bae KS. Evaluation of the pharmacokinetics of the DPP-4 inhibitor gemigliptin when coadministered with rosuvastatin or irbesartan to healthy subjects. Curr Med Res Opin. 2015 Feb;31(2):229-41. doi: 10.1185/03007995.2014.980886. Epub 2014 Nov 6. PMID 25350224